CLINICAL TRIAL: NCT02934737
Title: Role of Some Markers in the Progression of Diabetes in Obese Patients: a 8-year Observational Study
Brief Title: Role of markErs in the progreSsion of dIabeteS in Obese paTIeNts
Acronym: RESISTIN
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Other Study IDs: 20160004418
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Obese Patients
Keywords: Obesity; Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Progression of diabetes
  Other Names: Variations of biochemical parameters

SUMMARY:
Obese patients will be enrolled from 2006 to 2014. The progression of diabetes mellitus will be observed (if any). Anthropometric and biochemical parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (body mass index >/= 30 Kg/m2
* Normal blood glucose (glycemia < 100 mg/dl)

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Output patients with obesity
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Progression of diabetes | 8 years
  evaluation of glycemia during 8 years
Anthropometric parameters | 8 years
  Weight
Anthropometric parameters | 8 years
  Waist circumference; hip circumference; abdominal circumference
Markers of progression of diabetes | 8 years
  Adiponectin
Markers of progression of diabetes | 8 years
  Resistin

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Derosa, MD, PhD, FESC, Principal Investigator — University of Pavia

IPD SHARING:
Plan to Share IPD: No